CLINICAL TRIAL: NCT00506168
Title: Phase II Study of Irinotecan in Combination With Capecitabine in Previously Untreated Patients With Metastatic Colorectal Cancer
Brief Title: Study of Irinotecan & Capecitabine in Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study drugs are not covered anymore by insurance.
Sponsor: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-01-024
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Colorectal Neoplasms; Secondary; Drug Therapy, Combination
Keywords: Colorectal neoplasms; Secondary; Drug therapy, combination; Irinotecan; Capecitabine
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Irinotecan, Capecitabine

SUMMARY:
This study is to evaluate the efficacy and safety of combination chemotherapy with irinotecan and capecitabine in previously untreated metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a single center, single arm, open-label, phase II study to evaluate the efficacy and safety of combination chemotherapy with irinotecan and capecitabine in previously untreated metastatic colorectal cancer.

Patients younger then 65 will be treated with irinotecan 100 mg/m2 on day 1 and 8 and capecitabine 1,000mg/m2 twice daily from day 1 to 14 every 3 weeks.For patiens equal to or older then 65, doses of irinotecan and capecitabine will be reduced to 60 mg/m2 and 750 mg/2, respectively.

Response assessment will be performed every 3 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal cancer
* ECOG performance status 0-2
* Mesurable lesions
* No prior chemotherapyk or radiotherapy for metastatic disease. Prior radiotherapy is permitted if it was not administered to target lesions selected for this study and provided it has been completed at least 4 weeks before registration
* Adjuvnat chemo or radiotherapy was completed at least 6 months prior to start study treatment
* Adequate organ functions
* Expected survival is longer then 6 months
* Informed consent

Exclusion Criteria:

* Prior systemic chemotherapy for metastatic disease
* Prior treatment with oxaliplatin or irinotecan
* CNS metastases
* Uncontrolled or severe cardiovascular disease
* Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy
* Other malignancy within the past 3 years except cured non-melanomatous skin cancer or carcinoma in situ of the cervix
* Psychiatric disorder or uncontrolled seizure that would preclude compliance
* Pregnant, nursing women or patients with reproductive potential without contraception
* Patients receiving a concomitant treatment with drugs interacting with capecitabine such as flucytosine, phenytoin, or warfarin et al.
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known dihydropyrimidine dehydrogenase (DPD) deficiency
* Major surgery within 3 weeks prior to study treatment starts, or lack of complete recovery from the effects of major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2001-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Maximal response rate and toxicities | During treatment

SECONDARY OUTCOMES:
Progression-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hae Jung, M.D., Principal Investigator
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea